CLINICAL TRIAL: NCT00176488
Title: A Phase II Trial of Sequential Epirubicin/Vinorelbine in Patients With Advanced Breast Cancer
Brief Title: Epirubicin and Vinorelbine in Treating Patients With Stage II, Stage III, or Stage IV Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Competing studies
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000539565; P30CA072720 (NIH); CINJ 040302 (Other: Cancer Institute of New Jersey)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Epirubicin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sequential epirubicin/vinorelbine (Experimental): For patients with stage IIB (T3N0), IIIA, or IIIB breast cancer, epirubicin and vinorelbine will be administered for up to 5 cycles. For patients with stage IV breast cancer, epirubicin and vinorelbine will be administered as long as there is evidence of continued response or stable disease and no evidence of cardiac or other serious toxicities.
  Interventions: Drug: epirubicin; Drug: vinorelbine

INTERVENTIONS:
Drug: epirubicin — Epirubicin (100 mg/m2) will be given on Day 1
  Other Names: epirubicin hydrochloride
Drug: vinorelbine — Vinorelbine (18.75 mg/m2) will be given on Days 3 and 17.
  Other Names: vinorelbine ditartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epirubicin and vinorelbine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving epirubicin together with vinorelbine may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving epirubicin together with vinorelbine works in treating patients with stage II, stage III, or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the efficacy of sequential use of epirubicin hydrochloride followed by vinorelbine ditartrate in patients with stage IIB, IIIA, IIIB, or IV breast cancer.
* Measure the biological response to this regimen in sequential tumor biopsies and peripheral mononuclear cells from these patients.
* Correlate tumor response with changes in the gene expression of microtubule-associated protein 4.

OUTLINE: Patients receive epirubicin hydrochloride IV on day 1 and vinorelbine ditartrate IV over 6-10 minutes on days 3 and 17. Patients also receive filgrastim (G-CSF) subcutaneously on days 4-14 or pegfilgrastim IV on day 4.

For patients with stage IIB (T3, N0), IIIA, or IIIB disease, treatment repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity. For patients with stage IV disease, treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and after course 1 for research studies. Patients with accessible tumor for biopsy undergo sequential biopsies and core needle biopsies at baseline and after course 1. Tumor tissue samples are used for determination of p53 status by western blot analysis, immunohistochemistry, and DNA sequencing. Microtubule-associated protein 4, p53, and p21/WAF1 expression is analyzed by western blotting.

After completion of study treatment, patients are followed for 1 month.

PROJECTED ACCRUAL: A total of 46 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IIB (T3, N0), IIIA, IIIB, or IV breast carcinoma
* Original tumor must be available for analysis of p53 status
* Measurable disease, defined as any lesion that can be accurately measured in ≥ 1 dimension with longest diameter ≥ 20 mm using conventional techniques OR ≥ 10 mm with spiral CT scan

  * Stage IIIB disease will be assessed by clinical exam (monitoring skin changes as well as tumor size)
* No visceral crisis (lymphangitic pulmonary spread, or liver or marrow replacement sufficient to cause significant organ dysfunction)
* No untreated CNS metastases
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-2
* Life expectancy ≥ 8 weeks
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Bilirubin normal
* AST ≤ 3 times normal (≤ 5 times normal if liver metastases are present)
* Creatinine ≤ 1.5 mg/dL
* Ejection fraction ≥ lower limit of normal by MUGA scan or ECG
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception
* No other malignancy except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* No pre-existing disease (i.e., cardiac, pulmonary, neurologic, or other disease) that the investigator judges to be clinically significant
* No active infectious process, severe malnutrition, or intractable emesis

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* At least 3 weeks since prior radiotherapy
* At least 3 weeks since prior chemotherapy

  * Maximum prior doxorubicin hydrochloride dose must be ≤ 300 mg/m² OR equivalent anthracycline (epirubicin hydrochloride) dose must be ≤ 540 mg/m² OR calculated total anthracycline dose must be ≤ 540 mg/m² (determined as 1.8 times total doxorubicin hydrochloride dose plus epirubicin hydrochloride dose)
* No prior chemotherapy for metastatic disease
* Prior adjuvant chemotherapy, radiotherapy, and/or hormonal therapy for breast cancer allowed
* No concurrent radiotherapy except for brain metastases

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L. Toppmeyer, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Cancer Institute of New Jersey (a comprehensive cancer center) from June 2003 through May 2009.
Groups:
- Sequential Epirubicin/Vinorelbine: For patients with stage IIB (T3N0), IIIA, or IIIB breast cancer, epirubicin and vinorelbine will be administered for up to 5 cycles. For patients with stage IV breast cancer, epirubicin and vinorelbine will be administered as long as there is evidence of continued response or stable disease and no evidence of cardiac or other serious toxicities.
  epirubicin : Epirubicin (100 mg/m2) will be given on Day 1
  vinorelbine : Vinorelbine (18.75 mg/m2) will be given on Days 3 and 17.
  Beginning on cycle 1, patients will receive G-CSF (Neupogen) at a dose of 5 mcg/kg on Day 4 of treatment for 10 days OR pegfilgrastim (Neulasta) 6 mg on Day 4 of treatment.
Period: Overall Study
Arm/Group | Sequential Epirubicin/Vinorelbine
Started | 31
Completed | 30
Not Completed | 1
Not completed — Initiated Cycle 1 Day 1 only | 1

BASELINE CHARACTERISTICS:
Groups:
- Sequential Epirubicin/Vinorelbine: For patients with stage IIB (T3N0), IIIA, or IIIB breast cancer, epirubicin and vinorelbine will be administered for up to 5 cycles. For patients with stage IV breast cancer, epirubicin and vinorelbine will be administered as long as there is evidence of continued response or stable disease and no evidence of cardiac or other serious toxicities.
  epirubicin : Epirubicin (100 mg/m2) will be given on Day 1
  vinorelbine : Vinorelbine (18.75 mg/m2) will be given on Days 3 and 17.
Arm/Group | Sequential Epirubicin/Vinorelbine
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of the Sequential Use of a DNA Damaging Drug (Epirubicin) Followed by a Vinca Alkaloid (Vinorelbine) in the Treatment of Breast Cancer.
Time Frame: 10 years
Population: Study was closed prematurely and insufficient data was collected.
Arm/Group | Sequential Epirubicin/Vinorelbine
Number analyzed (Participants) | 0

2. Secondary Outcome: Biological Response to Epirubicin and Vinorelbine Administered in Patients With Breast Cancer in Sequential Tumor Biopsies and Peripheral Blood Mononuclear Cells.
Time Frame: 10 years
Population: Study was closed prematurely and insufficient data was collected.
Arm/Group | Sequential Epirubicin/Vinorelbine
Number analyzed (Participants) | 0

3. Secondary Outcome: Correlate Tumor Response With Changes in the Gene Expression of Microtubule Associated Protein 4 (MAP4).
Time Frame: 10 years
Population: Study was closed prematurely and insufficient data was collected.
Arm/Group | Sequential Epirubicin/Vinorelbine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 5 years and 6 months
Arm/Group | Sequential Epirubicin/Vinorelbine
Serious Adverse Events (participants affected / at risk) | 14/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequential Epirubicin/Vinorelbine (N=31)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 1 (1)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (General disorders) | 12 (14)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary-Other (Specify, malignant pleural effusion) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other Toxicity - Bilateral Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequential Epirubicin/Vinorelbine (N=31)
Alopecia (Skin and subcutaneous tissue disorders) | 29 (39)
Nail changes (Skin and subcutaneous tissue disorders) | 6 (6)
Dermatology/Skin-Other (Specify,_____) (Skin and subcutaneous tissue disorders) | 5 (6)
Bruising (in absence of grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 26 (48)
Constipation (Gastrointestinal disorders) | 15 (33)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 15 (24)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 13 (17)
Vomiting (Gastrointestinal disorders) | 10 (16)
Dyspepsia/heartburn (Gastrointestinal disorders) | 9 (13)
Anorexia (Gastrointestinal disorders) | 8 (14)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 7 (9)
Gastrointestinal-Other (Specify,_____) (Gastrointestinal disorders) | 3 (5)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 2 (5)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 25 (55)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 7 (7)
Pain-Other (Specify,___) (General disorders) | 18 (36)
Bone pain (General disorders) | 6 (6)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 5 (8)
Headache (General disorders) | 4 (5)
Abdominal pain or cramping (Gastrointestinal disorders) | 2 (3)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest pain (non-cardiac and non-pleuritic) (General disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 23 (68)
Platelets (Blood and lymphatic system disorders) | 11 (20)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 10 (27)
Blood/Bone Marrow-Other (Specify,_____) (Blood and lymphatic system disorders) | 4 (10)
Neuropathy-sensory (Nervous system disorders) | 10 (14)
Insomnia (Nervous system disorders) | 7 (7)
Dizziness/lightheadedness (Nervous system disorders) | 6 (9)
Mood alteration-anxiety, agitation (Psychiatric disorders) | 3 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 11 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Hyperglycemia (Investigations) | 6 (10)
Hypokalemia (Investigations) | 6 (8)
Hyponatremia (Investigations) | 4 (4)
Metabolic/Laboratory-Other (Specify,_____) (Investigations) | 4 (6)
Hypocalcemia (Investigations) | 3 (3)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (General disorders) | 9 (11)
Infection without neutropenia (Infections and infestations) | 2 (2)
Edema (Vascular disorders) | 9 (11)
Hypotension (Cardiac disorders) | 2 (2)
Alkaline phosphatase (Hepatobiliary disorders) | 7 (9)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 2 (3)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 2 (2)
Hot flashes/flushes (Endocrine disorders) | 4 (4)
Tearing (watery eyes) (Eye disorders) | 2 (2)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2)
Hemorrhage-Other (Specify,_____) (Blood and lymphatic system disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes